CLINICAL TRIAL: NCT02522611
Title: An Open-Label, Phase 1b Safety and Efficacy Trial of Periganglionic Resiniferatoxin for the Treatment of Intractable Pain Due to Cancer-induced Bone Pain
Brief Title: Periganglionic Resiniferatoxin for the Treatment of Intractable Pain Due to Cancer-induced Bone Pain
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150175; 15-N-0175
Record Dates: First submitted 2015-08-12; First posted 2015-08-13 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2025-09-09

CONDITIONS: Intractable Pain; Palliative Care
Keywords: Palliative Care; Adults; Cancer Pain; Quality of Life
MeSH Terms: conditions — Pain, Intractable; Cancer Pain | interventions — resiniferatoxin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Resiniferatoxin (Experimental): Schedule a maximum of 3 periganglionic DRG injection(s) at contiguous level(s) to treat targeted DRG responsible for chronic CIBP
  Interventions: Drug: Resiniferatoxin

INTERVENTIONS:
Drug: Resiniferatoxin — Resiniferatoxin (RTX) is an ultrapotent agonist analog of capsaicin that targets a receptor expressed on specific dorsal root sensory ganglia (DRG) neurons and is expected to reduce pain within the targeted zone.

SUMMARY:
Background:

Cancer-induced bone pain (CIBP) is common in people with cancer. Bone cancer can also lead to anxiety, depression, and reduced mobility and quality of life. Researchers believe a research drug called resiniferatoxin (RTX) may be able to help.

Objective:

To learn whether RTX is safe and can reduce cancer induced bone pain.

Eligibility:

People ages 18 and older with CIBP that is not relieved by standard treatments

Design:

Participants will have up to 6 outpatient visits over about 7 months. These will include:

Medical history

Physical exam

Blood and urine tests.

Thermal testing: a disk placed on the skin to test ability to sense temperature in and around the area of pain

Chest x-ray

EKG: stickers are placed on the chest to measure heart signals

ECG: measures electrical activity of the heart

Participants will have 1 inpatient visit lasting 2-4 days. This will include:

Catheter inserted into a vein in the arm. They are given anesthesia, sedation, and x-ray contrast.

A needle is passed through the skin of the back to inject the RTX.

Participants will keep a log of the pain medications they take after surgery.

Participants will be called 1 week and 2, 3, and 4 months after the injection.

Participants will be mailed surveys and questionnaires to complete 2, 3, and 4 months after the injection.

DETAILED DESCRIPTION:
Cancer-induced bone pain (CIBP) is a common clinical problem. While primary osteosarcoma is relatively uncommon, bone metastases frequently cause cancer-related pain with metastatic spread to bone in 60-84% of cases. Resiniferatoxin (RTX) is an ultrapotent agonist analog of capsaicin that targets a receptor expressed on specific dorsal root sensory ganglia (DRG) neurons and is expected to reduce pain within the targeted zone. The overall program goal is to develop a new treatment for intractable chronic pain below the mid-thoracic level resulting from CIBP that has not been controlled with conservative treatments.

Objectives:

The primary objective it to determine the maximum tolerated dose (MTD) of RTX when injected near one or more DRGs, to characterize its safety/toxicity profile, and to identify any dose-limiting toxicity (DLT). The secondary objectives are to determine the relative change in pain reduction, the change in opioid analgesic consumption and quality of life prior to RTX injection and at the various post RTX timepoints.

Study Population

Up to 30 adult subjects are estimated to be necessary for enrollment to have up to 16 subjects who will receive RTX and provide study-related assessment results through the 30-day time point.

Design

The study is a single center, open-label Phase 1b dose escalation safety and efficacy trial for adult subjects with intractable pain due to CIBP below the mid-thoracic level. Those subjects who meet all inclusion and exclusion criteria will undergo various study procedures and then be scheduled for the unilateral periganglionic (PG) DRG injection(s) (a maximum of 3 contiguous levels) under fluoroscopic guidance to treat the targeted DRGs demonstrated to be responsible for the chronic CIBP. The RTX will be injected at 1 of 4 dose levels, 0.8mcg/DRG, 1.6 mcg/DRG, 3.2 mcg/DRG or 6.4 mcg/DRG. The adaptivedesign algorithm for this study utilizes outcome dependent randomization, a process that selects the dose to be administered to the next subject based on all previous outcomes. In this schema, DLT is the measure that will be used to determine if it is safe to escalate to the next highest dose level.

Subjects who are screen failures and those who prematurely terminate participation will be replaced until 16 subjects have received the injection(s) and completed study-related assessments through the day 30 (D30) timepoint. There is no placebo group because of the invasive nature of the injection and the dose escalation performed in the study.

Outcome Measures

The primary outcome is to achieve a dose-response relationship for safety. All subjects will receive RTX. The secondary outcome measures are: 1) change in NRS and VAS scores at the post-RTX assessments compared to pre RTX assessment, 2) change of opioid usage (in MME) at post RTX assessments compared to pre RTX assessment; 3) comparison SF-36 and BDI at pre RTX injection and Days 14, 37, and 187.

The efficacy outcome variable will be evaluated by establishing dose-response curves, with dose plotted on the x-axis and changes in efficacy endpoints (before RTX treatment and at the post RTX assessment visits) plotted on the y-axis. If, at the end of the study, all dose levels of RTX have equal pain-relieving efficacy, the Data Safety Monitoring Committee (DSMC) may determine if it is appropriate to include a dose lower than 0.8 mcg and/or a control group. On the other hand, if the dose-response curves show that higher doses could result in greater pain-relieving efficacy, the protocol may be amended to include higher doses of RTX.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Male or female subjects must be at least 18 years of age or older.
2. Must be diagnosed with histologically-confirmed cancer-induced bone pain producing intractable chronic pain in the target area (mid thoracic or chest level down to lower extremities) which was poorly responsive to conservative therapies based on patient report, such as analgesic medication management with potent opioids with or without prior radiotherapy, bisphosphonates, or radioisotope therapy. Additionally, pain that is non-responsive to non-opioid drugs in situations where opioids were not tolerated. Conservative therapies do not include invasive treatments, such as neurolytic procedure, including surgical neurolysis, percutaneous regional or neuraxial continuous infusions (whether opioid or local anesthetic), and peripheral neuromodulation or spinal cord stimulation, but may include temporary diagnostic or therapeutic procedures.
3. Not currently seeking or receiving potentially curative therapies for cancer (e.g., chemotherapy or immunotherapy). Curative cancer therapy may be sought after the Outpatient Follow Up visit 14 (D14). Palliative anti-tumor therapy is allowed as long as the subject was established on that therapy prior to enrollment.
4. Must have moderate to severe pain that is not relieved by standard treatments. Mean daily worst pain NRS score of greater than or equal to 6 for pain at or below the T6 dermatome (level of the chest) that is associated with a malignant disease. The mean score must be derived from recordings on at least 4 of 7 consecutive days within 3 weeks preceding treatment.
5. The subject must agree to undergo a diagnostic periganglionic injection(s) with a long-acting local anesthetic (e.g., bupivacaine) under fluoroscopic guidance which resulted in at least a 30% temporary pain reduction in the targeted pain region lasting for the expected duration of the local anesthetic used.
6. Must be healthy enough to tolerate study procedures in the judgment of the investigator.
7. Subjects taking aspirin, non-steroidal anti-inflammatory medications, or vitamin supplements that include vitamin E or any prophylactic anticoagulant (including but not limited to Coumadin, heparin, or Xarelto) will be counseled either to stop taking these at least 7 days before surgery or be given instructions on dosing changes if applicable. In addition, if patients are currently taking a Factor Xa inhibitor (such as Xarelto) a hematology consult will be obtained. Subjects must be willing to comply with this requirement, which is standard clinical practice when undergoing elective surgical procedures to avoid surgical and post-surgical bleeding complications.
8. Formal review of the subject s medical records and written approval for his/her inclusion in the study by 3 separate persons:

   * Principal Investigator (PI) or an Associate Investigator (AI).
   * Medical oncologist or oncologic surgeon.
   * A member of the Pain and Palliative Care Service (PPCS) at the NIH.
9. For women of childbearing potential and men with partners of childbearing potential, the ability and willingness use an effective method of contraception during the study.

   Effective methods of birth control include:
   * hormonal contraception (birth control pills, injected hormones, or vaginal ring).,
   * intrauterine device.
   * barrier methods (condom or diaphragm) combined with spermicide
   * surgical sterilization (hysterectomy, tubal ligation, or vasectomy).
10. Medical clearance from referring physician consisting of a statement indicating an adequate recovery period from other previous trials/medication if known.
11. Must be able and willing to undergo an eye examination.
12. Must be able to read, speak and understand English and willing to complete the study tools and forms.
13. Subjects must have provided written informed consent which includes signing the institutional review board (IRB)-approved consent form prior to participating in any study-related activity.
14. Must have the capacity to provide informed consent.
15. Must have a responsible adult to provide assistance with activities of daily living as needed for the subject through the Day 14 visit.
16. Must have abilityAbility to assign a Durable Power of Attorney (DPA) for research and medical care at NIH.

EXCLUSION CRITERIA:

Subjects will be excluded from the study if they meet any of the following criteria:

1. Subject must not have primary pain source from anatomical regions at T5 dermatome or above.
2. Subject must not have pain due to causes other than cancer or its treatment that is moderate to severe in intensity.
3. Subjects must not be undergoing or have plans to undergo any active treatment for their cancer during the study until after the day 14 assessment timepoint, after the RTX injection.
4. Subject must not be anticipating initiation of palliative anti-tumor therapy or significant changes to current palliative anti-tumor therapy before completion of the Day 14 visit.
5. Subject must not have an ECG abnormality of which the baseline QTc interval exceeds 450 milliseconds.
6. Subjects must not have an allergy or hypersensitivity to chili peppers, capsaicin or radiographic contrast agents.
7. Subject must not have an anatomic abnormality or pathology of the spinal cord and/or PG space on magnetic resonance imaging (MRI) that could increase the risk of adverse effects of placement of the needle.
8. Subject must not have a contraindication to MRI or MRI contrast..
9. Subjects must not have evidence of a coagulopathy or hemostasis problem as

   evidenced by the following blood laboratory values within the week prior to the planned injection:
   * PT/INR (prothrombin time/International normalized ratio) > 1.5 times upper limit of normal range (ULN).
   * PTT (partial thromboplastin time) > 35 seconds.
10. Subjects must not have a platelet count <50,000/mm3. Platelets will be transfused as necessary to raise the platelet count to greater than or equal to 100,000/mm3 prior to dosing.
11. Subjects must not have a total neutrophil count (TNC) <1500. The US Clinical Practice Guideline for lumbar puncture is a platelet count of 50,0000, which is higher risk for hemorrhage than periganglionic infection. Patients with TNC<1500 (neutropenia) may be eligible later if their TNC level becomes greater than 1500 spontaneously or after use of medications stimulating granulocyte production, such as Neupogen (granulocyte colony stimulating factor: G-CSF).
12. Subjects must not have abnormal electrolyte levels (i.e. low potassium) that cannot be corrected.
13. Subjects must not be febrile or have other evidence of an infection within 7 days of the planned periganglionic injection.
14. Subjects must not have an allergy or hypersensitivity to chili peppers, capsaicin, or radiographic contrast agents.
15. Female subjects must not be pregnant or breastfeeding.
16. Subjects with any medical condition that, in the Investigator s opinion, could adversely impact the subject s participation or safety, conduct of the study, or interfere with the pain assessment, such as poorly controlled diabetes or hypertension. Patients can be re-assessed for eligibility if these conditions can be controlled medically.
17. Subjects may not have a history of heart failure or unexplained fainting (syncope).
18. Subjects may not have a known family history of long QT syndrome.
19. Subjects who participated in a clinical trial of an investigational drug or device within 30 days of screening visit or are scheduled to receive an investigational product within 14 days of RTX injection.
20. Subjects must not have received invasive treatments, such as a neurolytic procedure, including surgical neurolysis, percutaneous regional or neuraxial continuous infusions (whether opioid or local anesthetic), peripheral neuromodulation or spinal cord stimulation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the safety and efficacy of RTX administered intrathecally in subjects with severe refractory pain associated with advanced cancer along with ED100, the MTD, or the maximum dose administered, whichever is achieved first during dose... | Day 7, Day 15, Day 68, Day 188
  The primary study outcome measures are related to safety and toxicity of the investigational agent. The primary study outcome measures are: DLT MTD of RTX

SECONDARY OUTCOMES:
Improved pain relief through the 180-day time point compared to baseline | Completion of study
  The average of the daily worst NRS scores will be used throughout the study for post-injection visits.
Substantially reduced (20%) pain at the 30-, 60-. 90-, and 180-day post-treatment time points compared to the pain experienced at baseline | Completion of study
  The average of the daily worst NRS scores will be used throughout the study for post-injection visits.
Substantially reduced (20%) concomitant opioid analgesic consumption | Completion of study
  The average of the daily worst NRS scores will be used throughout the study for post-injection visits.
Improved quality of life | Completion of study
  The BPI is a validated tool designed to assess the severity of pain and the impact of pain on daily functions in patients with cancer pain and pain due to other chronic diseases.

CONTACTS AND LOCATIONS:
Overall Officials: John D Heiss, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do plan to share IPD. we will share all IPD that results in a publication on a public repository, as required by most journals. the data will be de-identified and anonymized.

REFERENCES:
- [Background] Mannes AJ, Brown DC, Keller J, Cordes L, Eckenhoff RG, Caudle RM, Iadarola MJ, Meng QC. Measurement of resiniferatoxin in serum samples by high-performance liquid chromatography. J Chromatogr B Analyt Technol Biomed Life Sci. 2005 Sep 5;823(2):184-8. doi: 10.1016/j.jchromb.2005.06.042. PMID 16039169
- [Background] Neubert JK, Mannes AJ, Karai LJ, Jenkins AC, Zawatski L, Abu-Asab M, Iadarola MJ. Perineural resiniferatoxin selectively inhibits inflammatory hyperalgesia. Mol Pain. 2008 Jan 16;4:3. doi: 10.1186/1744-8069-4-3. PMID 18199335
- [Background] Iadarola MJ, Mannes AJ. The vanilloid agonist resiniferatoxin for interventional-based pain control. Curr Top Med Chem. 2011;11(17):2171-9. doi: 10.2174/156802611796904942. PMID 21671877
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-N-0175.html